CLINICAL TRIAL: NCT01830374
Title: Weight Suppression, Dieting, and Bulimia Nervosa: A Biobehavioral Study
Brief Title: Bulimia Nervosa: A Biobehavioral Study (The Eating Disorder Study)
Acronym: TEDS
Status: Completed | Type: Observational
Sponsor: Drexel University (Other)
Collaborators: Columbia University (Other); The Miriam Hospital (Other)
Responsible Party: Principal Investigator, Michael Lowe, Professor, Drexel University
Other Study IDs: 12090001548
Record Dates: First submitted 2013-03-29; First posted 2013-04-12 (Estimated); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Bulimia Nervosa
Keywords: Bulimia nervosa; Eating disorder; Weight suppression; Dieting
MeSH Terms: conditions — Bulimia Nervosa; Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women with bulimia nervosa: This is not a treatment study. All participants will go through the same steps.

SUMMARY:
The purpose of this study is to examine biological (e.g., energy expenditure, neuroendocrine and appetitive hormones)and behavioral (e.g., binge eating and purging) correlates of weight suppression and current dieting status in women with bulimia nervosa. The investigators have differentiated between a diet-induced long-term energy imbalance (weight suppression, or the difference between one's highest-ever body weight and current weight) and a short-term energy imbalance (current dieting to either lose weight or avoid weight gain). This study will elucidate how two common yet largely unexplored types of dieting influence biological and behavioral variables in patients with bulimia nervosa, which could lead to modifications of prevailing models of bulimia nervosa and new strategies for improving treatment outcome.

DETAILED DESCRIPTION:
Bulimia nervosa (BN) is a debilitating psychiatric disorder that primarily affects young women. Empirically supported treatments for BN have been identified but less than half of treated individuals achieve long-term remission from the disorder, possibly because current treatment approaches do not sufficiently account for variables that help maintain the disorder. Psychosocial models of BN emphasize the role of dieting as a proximal cause of binge eating and purging. Dieting has both psychological and biological facets but existing models of BN have overwhelmingly focused on its psychological impact. The investigators have differentiated between a diet-induced long-term energy imbalance (weight suppression (WS), or the difference between one's highest-ever body weight and current weight) and a short-term energy imbalance (current dieting to either lose weight or avoid weight gain). Recent research has shown that WS levels in BN are elevated and that degree of WS predicts the severity of various BN characteristics and its clinical course. Studies of current dieting (CD) to lose weight have found that it is associated with reduced binge eating in BN, a finding that conflicts with prevailing models of the disorder. The proposed research will examine biological (e.g., energy expenditure, neuroendocrine and appetitive hormones) and behavioral (e.g., binge eating and purging) correlates of WS and CD in those with BN. (Relatively few of those with BN report dieting to avoid weight gain but its biological and behavioral correlates will also be examined.) The project will recruit 132 women (66 at Drexel University and 66 at Columbia University) meeting provisional Diagnostic and Statistical Manual-V diagnostic criteria for BN. The investigators will test the hypotheses that 1) CD and elevated WS will be associated with alterations in biological indices of metabolism and appetite, 2) WS will predict greater binge eating and purging, and CD will predict less binge eating, measured using Ecological Momentary Assessment (EMA), and 3) higher real time ratings of daily food restriction intentions will predict a reduced probability of binge eating during the same day but an increased probability of binge eating in subsequent days. Assessments for all participants will include: weight and reported previous highest weight (to calculate WS), the Eating Disorders Examination, 14 days of EMA to assess food restriction intentions, binge eating and purging episodes, three 24-hr food recalls, and resting energy expenditure and metabolic and appetitive hormones (including complete thyroid panel, leptin, ghrelin, cortisol and estradiol). Participants will be asked to return 6 months later for follow-up assessments of weight. This study will elucidate how two common yet largely unexplored types of dieting influence biological and behavioral variables in patients with BN, which could lead to modifications of prevailing models of BN and new strategies for improving treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bulimia nervosa according to the proposed DSM-V criteria
* Either currently receiving eating disorder treatment or actively seeking treatment
* BMI above 18.5 and below 30
* Not experiencing any signs of menopause
* Medically stable as determined by each site's study physician

Exclusion Criteria:

* Change in pharmacological treatment over past 4 weeks
* Currently taking atypical antipsychotic medications
* History of anorexia nervosa within the past year
* Pregnancy
* Currently taking medications that could alter hormone levels or metabolism
* Disorders affecting metabolism or hormone levels
* Non-removal metallic object
* Co-occurring severe mental illness
* At risk for suicide

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants will be recruited from local university counseling centers and eating disorder centers.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2012-08; Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Purging | 2 week EMA period
  Number of purging episodes recorded over two weeks.
Binge Eating | 2 week EMA period
  Number of binge eating episodes over two week period.
Hormone levels | Site Visit 3 (2 weeks)
  Hormone levels will be assessed approximately two weeks post-baseline at one time point.
Energy intake | Three weeks
  Energy intake (more specifically, energy density) will be assessed as an average of three dietary food recalls approximately three weeks post-baseline.
Resting metabolic rate (RMR) | Two weeks
  RMR will be assessed at Site Visit 3, approximately two weeks post-baseline.
Total percent body fat | Two weeks
  Total percent body fat will be assessed at Site Visit 3 (approximately 2 weeks post-baseline) using dual energy x-ray absorptiometry.

SECONDARY OUTCOMES:
Body weight | 6 months
  Body weight will be assessed at 6-month follow-up.
Psychosocial measures | Site Visit-Baseline
  Psychosocial self-report measures will be given at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Michael R. Lowe, Ph.D., Principal Investigator — Drexel University; Laurel Mayer, M.D., Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Columbia University, New York, New York
  - Drexel University, Philadelphia, Pennsylvania